CLINICAL TRIAL: NCT01672151
Title: Efficacy of Rapamycin Therapy With Chronic Immune Thrombocytopenia
Acronym: ITP
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Suzhou Medical College (Other)
Responsible Party: Principal Investigator, Zhaoyue Wang, Jiangsu Institute of hematology, First Affiliated Hospital of Suzhou Medical College
Other Study IDs: jsxys456
Record Dates: First submitted 2012-08-17; First posted 2012-08-24 (Estimated); Last update posted 2012-08-24 (Estimated); Status verified 2012-08

CONDITIONS: Immune Thrombocytopenic Purpura
Keywords: Refractory Immune Thrombocytopenic Purpura; rapamycin; regulatory T cells
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Sirolimus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: rapamycin — 4mg oral administration on the first day, 2 mg/d oral administration for 3 months
  Other Names: sirolimus

SUMMARY:
The aim of our study is to evaluate the efficacy of rapamycin with Refractory Immune Thrombocytopenic Purpura (RITP) and explore the further mechanism.

DETAILED DESCRIPTION:
Rapamycin, an immunosuppressive drug, is widely used to prevent allograft rejection and autoimmune diseases. Many studies have shown that the drug contributes to the expansion of regulatory T cells and preserves the highly suppressive function of autoreactive T cells. Patients with RITP often display a decreased proportion of regulatory T cells by flow cytometer, therefore, the investigators will examine the efficacy of rapamycin in RITP patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnoses of idiopathic thrombocytopenic purpura
* Hormone and immune suppression, splenectomy is invalid

Exclusion Criteria:

* patients had a bad tolerance to rapamycin
* platelet counts < 10*10E9/L during the treatment of rapamycin

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 35 patients using rapamycin therapy were observed before and after treatment,who did not response to any other administrations including prednisone and immunosuppressive drugs, even splenectomy .
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2011-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: zhaoyue wang, doctor, Study Director
Locations (1):
- Jiangsu Institute of Hematology, Suzhou, Jiangsu, China